CLINICAL TRIAL: NCT02280525
Title: A Study of Umbilical Cord Blood-Derived Natural Killer Cells in Conjunction With Lymphodepleting Chemotherapy and Lenalidomide as Immunotherapy in Patients With Hematologic Malignancies
Brief Title: Cord Blood Natural Killer (NK) Cells in Leukemia/Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0297; P-TRP-1996-14 (Other Grant/Funding Number: Leukemia & Lymphoma Society (LLS)); NCI-2014-02678 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic Lymphocytic Leukemia; CLL; Natural Killer Cells; NK; Umbilical Cord Blood; UCB; Lenalidomide; CC-5013; Revlimid; Rituximab; Rituxan; Fludarabine; Fludarabine phosphate; Fludara; Cyclophosphamide; Cytoxan; Neosar; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Rituximab; fludarabine; fludarabine phosphate; Cyclophosphamide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lymphodepleting Chemotherapy Option #1 (Experimental): Preferred regimen for CLL and low grade lymphoma
  Lenalidomide 2.5 mg by mouth once a day on Days -2 through Day +14. Fludarabine 25 mg/m2 by vein over 1 hour on Days -5 to -3. Cyclophosphamide 200 mg/m2 by vein over 3 hours on Days -5 to -3. Rituximab 375 mg/m2 by vein over 3-6 hours on Day -5 for participants with B-cell cancer.
  Dose Escalation Phase Starting Dose Level of NK Cells: 1 x 10^7 NK cells/kg given by vein on Day 0.
  Dose Expansion Phase Starting Dose level of NK cells: Maximum tolerated dose from Dose Escalation Phase.
  Interventions: Drug: Lenalidomide; Drug: Rituximab; Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: NK Cells
- Lymphodepleting Chemotherapy Option #2 (Experimental): For all malignancies if able to tolerate higher dose cyclophosphamide per the discretion of the treating physician
  Lenalidomide 2.5 mg by mouth once a day on Days -2 through Day +14. Fludarabine 25 mg/m2 by vein over 1 hour on Day -6 to -2. Cyclophosphamide 60 mg/kg by vein over 3 hours on Days -5 and -4.
  Dose Escalation Phase Starting Dose Level of NK Cells: 1 x 10^7 NK cells/kg given by vein on Day 0.
  Dose Expansion Phase Starting Dose level of NK cells: Maximum tolerated dose from Dose Escalation Phase.
  Interventions: Drug: Lenalidomide; Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: NK Cells
- Lymphodepleting Chemotherapy Option #3 (Experimental): For myeloid malignancies
  Lenalidomide 2.5 mg by mouth once a day on Days -2 to Day +14. Fludarabine 30 mg/m2 by vein over 1 hour on Days -6 to -2. Cytarabine 2 mg/m2 by vein on Days -6 to -2.
  Dose Escalation Phase Starting Dose Level of NK Cells: 1 x 10^7 NK cells/kg given by vein on Day 0.
  Dose Expansion Phase Starting Dose level of NK cells: Maximum tolerated dose from Dose Escalation Phase.
  Interventions: Drug: Lenalidomide; Drug: Fludarabine; Procedure: NK Cells; Drug: Cytarabine

INTERVENTIONS:
Drug: Lenalidomide — 2.5 mg by mouth daily on Day -2 to Day +14.
  Other Names: CC-5013; Revlimid
Drug: Rituximab — 375 mg/m2 by vein on Day -5 for participants with B-cell cancer.
  Other Names: Rituxan
  Arms: Lymphodepleting Chemotherapy Option #1
Drug: Fludarabine — Lymphodepleting Chemotherapy Option #1: Fludarabine 25 mg/m2 by vein on Days -5 to -3.
  Lymphodepleting Chemotherapy Option #2: Fludarabine 25 mg/m2 by vein over 1 hour on Day -6 to -2.
  Lymphodepleting Chemotherapy Option #3: Fludarabine 30 mg/m2 by vein over 1 hour on Days -6 to -2
  Other Names: Fludarabine Phosphate; Fludara
Drug: Cyclophosphamide — Lymphodepleting Chemotherapy Option #1: Cyclophosphamide 200 mg/m2 by vein on Days -5 to -3.
  Lymphodepleting Chemotherapy Option #2: Cyclophosphamide 60 mg/kg by vein over 3 hours on Days -5 and -4.
  Other Names: Cytoxan; Neosar
  Arms: Lymphodepleting Chemotherapy Option #1; Lymphodepleting Chemotherapy Option #2
Procedure: NK Cells — Participant assigned to a dose level of NK cells based on when joined study. Starting dose level of NK cells 1 x 10^7 NK cells/kg given by vein on Day 0.
  NK Cell Infusion Expansion Phase: Maximum tolerated dose of NK cells from Induction Phase.
Drug: Cytarabine — Cytarabine 2 mg/m2 by vein on Days -6 to -2.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
  Arms: Lymphodepleting Chemotherapy Option #3

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of immune cells called natural killer (NK) cells that can be given with chemotherapy to patients with CLL. Researchers want to learn if adding NK cells will be effective in treating the disease. The safety of this will also be studied.

NK cells may kill cancer cells that remain in your body after your last chemotherapy treatment. The NK cells will be separated from umbilical cord blood. The device used in the laboratory to separate the NK cells is called a CliniMACS. These separated NK cells will then be grown in the lab to increase the number of NK cells that can be given to you by vein.

This is an investigational study. Rituximab, fludarabine, and cyclophosphamide are FDA approved and commercially available for the treatment of CLL. Cytarabine, filgrastim, and lenalidomide are FDA approved and commercially available for the treatment of other types of cancer. The use of cytarabine, filgrastim, and lenalidomide for the treatment of CLL is investigational.

The use of NK cells is investigational. The NK cell process is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 44 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Central Venous Catheter:

The chemotherapy, some of the other drugs in this study, and the NK cells will be given by vein through your central venous catheter (CVC). A CVC is a sterile flexible tube and needle that will be placed into a large vein while you are under local anesthesia. Blood samples will also be drawn through your CVC. The CVC will remain in your body during treatment. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

NK Cell Dose Levels:

You will be assigned to a dose level of NK cells based on when you joined this study. Up to 5 dose levels of NK cells will be tested. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of NK cells is found.

If not enough NK cells can be produced in the laboratory for your assigned dose level, you will still receive the NK cells that were produced. If you are infused with a lower number of NK cells than had been originally planned, the CLL may not respond. Researchers do not know what number of NK cells is needed for a response.

Chemotherapy and NK Cell infusion:

The days before you receive the NK cells are called minus days. The day you receive the NK cells is called Day 0. The days after you receive the NK cells are called plus days.

You will receive 1 of 3 study drug plans. Your doctor will decide which plan you will receive based on your age, prior treatment, diagnosis, and health status. You will receive 1 of the 3 options as explained below.

Option #1:

On Day -2 through Day +14, you will take lenalidomide by mouth once a day at about the same time each day. If you are able to do so, you will take aspirin or another drug as instructed by your doctor on these days to help prevent blood clots. You will be asked to complete a study drug diary and bring it to each study visit. The study staff will tell you more about this.

On Day -5, you will receive fludarabine by vein over 1 hour and cyclophosphamide by vein over 3 hours. If you have a B-cell cancer, you will receive rituximab by vein over 3-6 hours. Rituximab and fludarabine are given to treat the cancer and lower the immune system in order to lower the risk of the body rejecting the NK cells. Cyclophosphamide is given to lower the immune system in order to lower the risk of graft-versus-host disease (GVHD -- when transplanted immune tissue, such as cord blood NK cells, attacks the tissues of the recipient's body).

On Day -4 and -3, you will receive fludarabine by vein over 1 hour and cyclophosphamide by vein over 3 hours.

On Days -2 and -1, you will rest.

On Day 0, you will receive NK cells by vein.

Option #2:

On Day -2 through Day +14, you will take lenalidomide by mouth once a day at about the same time each day. If you are able to do so, you will take aspirin or another drug as instructed by your doctor on these days to help prevent blood clots. You will be asked to complete a study drug diary and bring it to each study visit. The study staff will tell you more about this.

On Day -6, you will receive fludarabine by vein over 1 hour. Fludarabine is given to treat the cancer and lower the immune system in order to lower the risk of the body rejecting the NK cells.

On Day -5, and -4, you will receive fludarabine by vein over 1 hour and cyclophosphamide by vein over 3 hours. Cyclophosphamide is given to lower the immune system in order to lower the risk of graft-versus-host disease (GVHD -- when transplanted immune tissue, such as cord blood NK cells, attacks the tissues of the recipient's body).

On Day -3 and -2, you will receive fludarabine by vein over 1 hour. Fludarabine is given to treat the cancer and lower the immune system in order to lower the risk of the body rejecting the NK cells.

On Day -1, you will rest.

On Day 0, you will receive NK cells by vein.

Option #3:

On Day -7, you be given fluids by vein to hydrate you.

On Days -6 through - 2, you will receive fludarabine by vein over 1 hour and cytarabine by vein over 1 hour.

On Day -2 through Day +14, you will take lenalidomide by mouth once a day at about the same time each day. If you are able to do so, you will take aspirin or another drug as instructed by your doctor on these days to help prevent blood clots. You will be asked to complete a study drug diary and bring it to each study visit. The study staff will tell you more about this.

On Day -1, you will rest.

On Day 0, you will receive NK cells by vein.

Starting on Day +5, you will receive filgrastim as an injection under the skin 1 time a day until your blood cell levels return to normal. Filgrastim is designed to help with the growth of white blood cells.

Study Visits:

Within 7 days before starting chemotherapy:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.

Within 2 days and then about 1 week, 2 weeks, 3 weeks, 1 month, 2 months, 3 months, and 4 months after the NK cell infusion, the following tests and procedures will be performed:

°Blood (about 4 tablespoons) will be drawn for routine tests, tests to measure levels of certain proteins, to learn how your body's immune system responds to the NK cell infusion, and to check the level of the NK cells.

About 1 week, 3 weeks, 1 month, and 4 months after the NK cell infusion, you will have a bone marrow biopsy/aspiration to check the status of the disease. To collect a bone marrow biopsy/aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone and bone marrow is withdrawn through a large needle.

Pregnancy Tests:

If you can become pregnant, blood (about 1 teaspoon each time) will be drawn for a pregnancy test within 10-14 days and 24 hours before you are prescribed lenalidomide, at about Day +21, at 2 months after NK cell infusion, and then again 4 weeks after therapy is stopped. To continue on this study, you must not be pregnant.

If possible, the blood needed for pregnancy tests will be collected during the above blood draws so that no additional needle sticks will be needed.

Length of Study:

You will be on study for up to about 1 year. You may be taken off study early if the disease gets worse, if you are unable to receive the NK cell infusion, if you have any intolerable side effects, if you are unable to follow study directions, if your doctor thinks it is in your best interest, if the study is stopped, or if you choose to leave the study early.

You should talk to the study doctor if you want to leave the study early. If you are taken off study early, you still may need to return for routine post-transplant follow-up visits, if your doctor decides it is needed.

If you are thinking about dropping out of this study, please tell the study doctor. The doctor can tell you about the effects of stopping treatment. You and the doctor can talk about what follow-up care and testing would help you the most.

If you leave the study, your test results and information cannot be removed from the study records.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of hematologic malignancies who have received at least 2 lines of standard chemoimmunotherapy and have persistent disease.
2. Patients with acute lymphoblastic leukemia (ALL), acute myelogenous leukemia (AML), chronic myelogenous leukemia (CML) with relapsed or refractory disease who are not eligible for stem cell transplantation or other standard therapies.
3. Patients with histologically confirmed aggressive hematologic malignancies with chemotherapy-refractory disease. Chemotherapy refractory disease is defined as one or more of the following: Stable disease or progressive disease as best response to most recent chemotherapy containing regimen or disease progression or recurrence within 12 months of prior Autologous or allogeneic stem cell transplant. Subjects must have received adequate prior therapy including at a minimum: anti-CD20 monoclonal antibody unless tumor is CD20-negative, an anthracycline containing chemotherapy regimen. Subjects with transformed FL must have received prior chemotherapy for follicular lymphoma and subsequently have chemo-refractory disease after transformation to diffuse large B-cell lymphoma (DLBCL).
4. Patient with Hodgkin's Lymphoma with relapsed or refractory disease who are not eligible for stem cell transplantation or other standard therapies.
5. Patients at least 3 weeks from last cytotoxic chemotherapy. Patients may continue tyrosine kinase inhibitors and/or lenalidomide until the day of study consent.
6. Karnofsky Performance Scale > 60%.
7. Adequate hepatic function, as defined by SGPT <3 X upper limit of normal; serum bilirubin and alkaline phosphatase <2 X upper limit of normal, or considered not clinically significant by the study doctor or designee, serum creatinine of </=2 mg/dl.
8. Able to provide written informed consent.
9. 18-80 years of age.
10. All study participants must be registered into the mandatory Revlimid REMSTM program, and be willing and able to comply with the requirements of the Revlimid REMSTM program. Females of childbearing potential must adhere to the scheduled pregnancy testing and contraception as required in the Revlimid REMSTM program. A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
11. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy.
12. Patients must have a CB unit available which is matched with the patient at 3, 4, 5, or 6/6 HLA class I (serological) and II (molecular) antigens.
13. Patients who are HIV positive must be willing to comply with effective antiretroviral therapy.

Exclusion Criteria:

1. Positive beta HCG in female of child-bearing potential defined as not postmenopausal for 24 months or no previous surgical sterilization or lactating females.
2. Presence of Grade 3 or greater toxicity from the previous treatment.
3. Concomitant use of other investigational agents.
4. Not consenting to participate in LAB00-099.
5. Patients with known hypersensitivity to lenalidomide and/or rituximab (CD20+ patients only).
6. Patients who are HIV positive with a detectable viral load > 750 copies/ml on adequate retroviral therapy must be evaluated for HIV drug resistance test (HIV-1 genotype). These patients may be enrolled only after discussion with the PI and the Infectious Disease team.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Natural Killer (NK) Cells with Lenalidomide and Lymphodepleting Chemotherapy | 30 days
  Primary objective is to determine maximum tolerated dose (MTD). Dose-limiting toxicity (DLT) target rate is at most 20%. DLT includes any grade 4 toxicity related to NK infusion related toxicity; grades 3-5 allergic reactions related to study cell infusion; grades 3-5 organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic) not pre-existing or due to underlying malignancy or due to preparative chemotherapy and occurring within 30 days post-NK infusion.

SECONDARY OUTCOMES:
Response Rate of Natural Killer (NK) Cells with Lenalidomide and Lymphodepleting Chemotherapy Determined by Bone Marrow Biopsy/Aspiration | 1 week, 3 weeks, 1 month, and 4 months after the NK cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org